CLINICAL TRIAL: NCT05170763
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics of Single Dose and 7-day Repeat Doses of PA9159 Nasal Spray in Healthy Chinese Adult
Brief Title: Safety, Tolerability, and Pharmacokinetics of PA9159 Nasal Spray in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA9159-101
Record Dates: First submitted 2021-09-28; First posted 2021-12-28 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Arm 1-4, the treatment is given once for one day, with escalation doses of 10 μg, 20 μg, 40 μg, 80 μg. Arm 5-6, PA9159 at the escalation dose of 20 μg and 40 μg is given once a day for 7 days. 10 health subjects will be enrolled for each dose group, randomized proportionally at 4:1 ratio to receive either the investigational product PA9159 or placebo nasal spray, with a total of 60 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled dose escalation phase 1 trial, including single dose and 7-day repeat doses of PA9159 nasal spray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PA9159 10 μg single dose and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either single dose of 10 μg PA9159 or placebo. There will be a one week follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 10 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 20 μg single dose and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either single dose of 20 μg PA9159 or placebo. There will be a one week follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 20 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 40 μg single dose and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either single dose of 40 μg PA9159 or placebo. There will be a one week follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 40 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 80 μg single dose and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either single dose of 80 μg PA9159 or placebo. There will be a one week follow-up period to review all available clinical and laboratory safety data.
  Interventions: Drug: PA9159 nasal spray solution, 80 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 20 μg repeated doses and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either 20 μg PA9159 or placebo once a day for 7 days. There will be a one week follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 20 μg 7-day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 40 μg repeated doses and placebo (Experimental): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either 40 μg PA9159 or placebo once a day for 7 days. There will be a one week follow-up period to review all available clinical and laboratory safety data.
  Interventions: Drug: PA9159 nasal spray solution, 40 μg 7-day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient

INTERVENTIONS:
Drug: PA9159 nasal spray solution, 10 μg one day treatment — Single dose of PA9159 (5 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, one spray each in the left and right nostril.
  Arms: PA9159 10 μg single dose and placebo
Drug: PA9159 nasal spray solution, 20 μg one day treatment — Single dose of PA9159 (5 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 20 μg single dose and placebo
Drug: PA9159 nasal spray solution, 40 μg one day treatment — Single dose of PA9159 (10 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 40 μg single dose and placebo
Drug: PA9159 nasal spray solution, 80 μg one day treatment — Single dose of PA9159 (10 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, four sprays each in the left and right nostril.
  Arms: PA9159 80 μg single dose and placebo
Drug: PA9159 nasal spray solution, 20 μg 7-day treatment — Repeated doses of PA9159 (5 μg/nasal spray) or Placebo is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 20 μg repeated doses and placebo
Drug: PA9159 nasal spray solution, 40 μg 7-day treatment — Repeated doses of PA9159 (10 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 40 μg repeated doses and placebo
Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient — Placebo is delivered intranasally through a metered-dose mechanical spray pump with the same volume as the corresponding PA9159 dose group

SUMMARY:
PA9159 is a highly potent novel corticosteroid. The purpose of this study is to exam the safety, tolerability, and pharmacokinetics of single and repeat dosing of intranasal PA9159, to establish maximum tolerated dose in healthy chinese adult

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled dose escalation phase 1 trial, including single dose and 7-day repeat doses of PA9159 nasal spray. In the first part of the study, the treatment is given once for one day, with escalation doses of 10 μg, 20 μg, 40 μg, 80 μg. In the second part of the study, PA9159 at the escalation dose of 20 μg and 40 μg is given once a day for 7 days. 10 health subjects will be enrolled for each dose group, randomized proportionally at 4:1 ratio to receive either the investigational product PA9159 or placebo nasal spray, with a total of 60 subjects for this two-part study. Subjects will be evaluated for the safety, tolerability and pharmacokinetics of PA9159 intranasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 65 years (including upper and lower limits);
* Male body weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 28 kg/m2 (including cut-off values);
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Those with a history or current history of serious diseases such as respiratory, cardiovascular, digestive, endocrine, hematological, immune, psychiatric, neurological, and otologic diseases, with special attention to a history of recurrent (defined as > 1) or disseminated herpes zoster, history of recurrent infections, tuberculosis infection, glaucoma and cataract; Suffering from acute, chronic or local infectious diseases (e.g., eye, nose infection, etc.);
* Those who are allergic to the study drug or any component of the study drug (refer to the susceptibility of the body to allergic reactions, or to a variety of food, drugs, or environmental substances);
* Any past or current medical history that may affect the safety of the study in the body, especially any nasal disorder affecting drug absorption: a) History of long-term nasal congestion, rhinorrhea, nasal pruritus, headache, epistaxis, etc.; b) asthma, aspirin stress response, chronic respiratory disease, etc.; c) History of nasal surgery, trauma, allergic rhinitis, chronic rhinitis, sinusitis, severe deviation of nasal septum, etc., and the researchers believe that it is still clinically significant;
* Abnormal and clinically significant vital signs, physical examination, nasal examination, laboratory tests (hematology, blood chemistry, urinalysis, coagulation function, serum cortisol), ECG, etc., during screening;
* Positive test results and have clinical significance for human immunodeficiency virus HIV-P24 antigen/antibody, hepatitis C virus (HCV) antibody, treponema pallidum (TP), or hepatitis B five items (hepatitis B surface antigen, hepatitis B surface antibody, hepatitis B e antigen, hepatitis B e antibody, and hepatitis B core antibody);
* Regular drinkers within 6 months prior to screening,That is, drink more than 14 units of alcohol per week (1 unit = 360 mL of beer containing 5% alcohol or 45 mL of spirits with 40% alcohol or 150 mL of wine with 12% alcohol content) or who have a positive alcohol breath test at screening or who cannot stop alcohol intake during the study;
* Smoking more than 5 cigarettes per day on average within 3 months prior to screening, or unable to discontinue the use of any tobacco products during the trial;
* History of drug abuse, history of drug abuse, or positive urine screening for drug abuse (including morphine, methamphetamine, ketamine, dimethyldioxymethamphetamine, tetrahydrocannabinol acid);
* Those who have taken any drugs (prescription drugs, over-the-counter drugs, Chinese herbal medicines, vaccines) or health products within 2 weeks prior to screening and during screening;
* Those who have used glucocorticoid-containing preparations or any drugs that affect CYP3A4 enzyme activity (e.g., ritonavir or ketoconazole, etc.) within 30 days prior to screening and during screening;
* Consumption of beverages or foods containing grapefruit, dragon fruit, mango, grapefruit, pomegranate, papaya, carambola within 14 days prior to screening and during screening, or who do not agree to stop eating the above-mentioned diet during the study;
* Consumption of any caffeine- and xanthine-rich food or beverages (coffee, tea, cola, chocolate, seafood, animal liver, etc.) within 48 hours prior to the first dose of study drug, or who do not agree to stop eating these diets during the study;
* It cannot be guaranteed that effective contraceptive measures or fertility planners or sperm or egg donors are taken during the trial and for at least 1 year after the last dose;
* Donation or massive blood loss (≥ 300 mL, except during female physiology) or use of blood products or transfusions within 90 days prior to screening and during screening;
* Participating in other clinical investigators or subjects participating in other clinical trials within 90 days prior to screening for less than 7 days;
* Major surgery (as judged by the investigator based on past medical history data), major trauma, or planned surgery during the study within 6 months prior to screening;
* Difficulty in venous blood collection, or a known history of multiple needle sickness and blood sickness;
* Women with a positive pregnancy test or breastfeeding;
* Other conditions that, in the opinion of the investigator, are not suitable for participation in the study or the subject is unable to participate in the study due to his/her own reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events (AEs) | up to 7 days after last nasal spray treatment
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Number of subjects having abnormal hematology laboratory parameters | within 24 hours after last nasal spray treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal clinical chemistry parameters | within 24 hours after last nasal spray treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal values for urinalysis | within 24 hours after last nasal spray treatment
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Body temperature | up to 24 hours after last nasal spray treatment
  Vital sign-Body temperature
Systolic and diastolic blood pressure | up to 24 hours after last nasal spray treatment
  Vital sign-Systolic and diastolic blood pressure
Pulse rate | up to 24 hours after last nasal spray treatment
  Vital sign-Pulse rate
ECG parameter-QTc interval | up to 24 hours after last nasal spray treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically calculates the QTc intervals
ECG parameter-PR interval | up to 24 hours after last nasal spray treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures PR intervals
ECG parameter-QRS duration | up to 24 hours after last nasal spray treatment
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QRS duration
Numbers of subjects experiencing local nasal/throat irritation symptoms | up to 24 hours after nasal spray treatment
  Self reported local irritation symptoms including pruritus, dryness, sneezing, nasal congestion, rhinorrhea, dry cough and odynophagia
Numbers of subjects showing signs of local reactions | up to 24 hours after nasal spray treatment
  Visual nasal examination will be conducted by a trained physician for presence of nasal cavity erythema, edema, epistaxis, perforation of the nasal septum, or any abnormal finding deemed clinically significant.

SECONDARY OUTCOMES:
Serum cortisol levels | From pre-dose until 24 hours post-dose
  Monitor the concentration changes of serum cortisol before and after PA9159 administration.
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-Cmax | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 10, 20, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-Tmax | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 10, 20, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-AUC | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 10, 20, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Area Under the Plasma Concentration-Time Curve (AUC)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-T1/2 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 10, 20, 30 minutes, 1, 1.5, 2, 3 , 4, 6, 8,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Half-Life Period (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing TongRen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No